CLINICAL TRIAL: NCT03878264
Title: An Open-label, 2-part Study Designed to Assess the Absolute Bioavailability of CORT118335 and Determine the Mass Balance Recovery, Absorption, Metabolism and Elimination, and Metabolite Profile and Identification of Metabolite Structures of [14C]-CORT118335 in Healthy Male Subjects
Brief Title: Absolute Bioavailability and Metabolism Study of CORT118335 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CORT118335-851; 2018-001507-36 (EudraCT Number)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — CORT118335

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): On Day 1, participants will receive a single oral dose of CORT118335 900 mg (Treatment A) after an overnight fast, and a 15-minute intravenous infusion of a microdose of 14C-CORT118335 (Treatment B) beginning 2 hours 45 minutes after the oral dose is administered.
  Interventions: Drug: CORT118335 Oral; Drug: 14C-CORT118335 intravenous
- Part 2 (Experimental): On Day 1, participants will receive a single oral dose of 14C-CORT118335 150 mg (Treatment C) after an overnight fast.
  Interventions: Drug: 14C-CORT118335 oral

INTERVENTIONS:
Drug: CORT118335 Oral — CORT118335 900 mg spray-dried dispersion in bottle and vehicle for oral administration
  Other Names: Treatment A
  Arms: Part 1
Drug: 14C-CORT118335 intravenous — 14C-CORT118335 solution for infusion 100 µg containing not more than 37 kiloBequerel (1 µCi) 14C
  Other Names: Treatment B
  Arms: Part 1
Drug: 14C-CORT118335 oral — 14C-CORT118335 oral solution 150 mg containing not more than 3.3 megaBequerel (90 µCi) 14C
  Other Names: Treatment C
  Arms: Part 2

SUMMARY:
This study will evaluate the absolute bioavailability of CORT118335 and determine the mass balance recovery, absorption, metabolism and elimination, and metabolite profile and identification of metabolite structures following a single oral dose of CORT118335 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age for Part 1 and 30 to 65 years of age for Part 2
* Body mass index of 18.0 to 30.0 kg/m^2
* Provide written informed consent
* Have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day) for Part 2
* Adhere to the contraception requirements.

Exclusion Criteria:

* Have received any investigational medicine in a clinical research study within the previous 3 months or CORT118335 at any time
* Employees or immediate family members of employees of the study site or Sponsor
* Have a pregnant partner
* History of abuse of any drug or alcohol, or regularly consume more than 21 units alcohol/week
* Smokers or users of e-cigarettes and nicotine replacement products within the last 6 months
* Occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017; greater than background radiation exposure from other sources exceeding 5 milliSieverts (mSv) in the last 12 months or 10 mSv in the last 5 years
* Clinically significant abnormal results of clinical laboratory safety tests, electrocardiogram, or measurement of heart rate and blood pressure
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, neurological, or gastrointestinal disease
* History and/or symptoms of adrenal insufficiency or any condition that could be aggravated by glucocorticoid blockade (e.g., an autoimmune disease; allergy requiring treatment)
* Donation or loss of greater than 400 mL of blood within the past 3 months
* Has consumed liquorice or other glycyrrhetic acid derivatives regularly in the past 6 months
* Are taking, or have taken, any prescribed, over-the-counter drug or vitamins/herbal remedies within 14 days (longer restrictions apply for some medicines).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-03-24 (Actual)

PRIMARY OUTCOMES:
Absolute Oral Bioavailability (F) of CORT118335 | Predose and at pre-specified time points up to Day 12
Mass Balance Recovery in Excreta After a Single Oral Dose of 14C-CORT118335 | Until the mass balance criteria have been met by all participants (estimated Day 17)
Mass Balance Recovery in Urine After a Single Oral Dose of 14C-CORT118335 | Until the mass balance criteria have been met by all participants (estimated Day 17)
Mass Balance Recovery in Feces After a Single Oral Dose of 14C-CORT118335 | Until the mass balance criteria have been met by all participants (estimated Day 17)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of Total Radioactivity after Oral Dosing: Peak Plasma Concentration (Cmax) | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Total Radioactivity in Plasma after Oral Dosing: Time from Dosing to Cmax (tmax) | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Total Radioactivity after Oral Dosing: Area Under the Plasma Concentration-time Curve from Zero Time to Time of the Last Measurable Concentration (AUC0-last) | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Total Radioactivity in Plasma after Oral Dosing: Apparent Elimination Half-life (t1/2) | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Total Radioactivity in Plasma after Oral Dosing: Mean Residence Time (MRT) | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Plasma CORT118335 after Oral Dosing: Cmax | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Plasma CORT118335 after Oral Dosing: Tmax | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Plasma CORT118335 after Oral Dosing: AUC0-last | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Plasma CORT118335 after Oral Dosing: MRT | Pre-dose and at pre-specified time points up to Day 15 after dosing
PK of Plasma 14C-CORT118335 after IV Dosing: Cmax | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Plasma 14C-CORT118335 after IV Dosing: AUC0-last | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Plasma 14C-CORT118335 after IV Dosing: t1/2 | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Plasma 14C-CORT118335 after IV Dosing: Total Clearance (CL) | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Plasma 14C-CORT118335 after IV Dosing: MRT | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Total Radioactivity in Plasma after IV Dosing: Cmax | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Total Radioactivity in Plasma after IV Dosing: AUC0-last | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Total Radioactivity in Plasma after IV Dosing: t1/2 | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Total Radioactivity in Plasma after IV Dosing: CL | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK of Total Radioactivity in Plasma after IV Dosing: MRT | Pre-dose and at pre-specified time points up to Day 12 after dosing
PK in Plasma after IV Dosing: AUC0-last for 14C-CORT118335 / AUC0-last for Total Radioactivity | Pre-dose and at pre-specified time points up to Day 12 after dosing
Distribution of Total Radioactivity into Red Blood Cells after Oral Dosing | Pre-dose and at pre-specified time points up to Day 15 after dosing
Number of CORT118335 Metabolites Accounting for >10% of Total Radioactivity Detected in Plasma, Urine, and Feces | Until the mass balance criteria have been met by all participants (estimated Day 17)
Percentage of Participants with One or More Adverse Events | Until the mass balance criteria have been met by all participants (estimated Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No